CLINICAL TRIAL: NCT06274333
Title: The Effect of Adding Dexmedetomidine or Tramadol to Paracetamol- An Effort to Attenuate Catheter Related Bladder Discomfort: A Randomized, Triple-Blind Clinical Trial
Brief Title: Adding Dexmedetomidine or Tramadol to Paracetamol- An Effort to Attenuate Catheter Related Bladder Discomfort
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Neveen Abd El Maksoad Kohaf, Lecturer of Clinical Pharmacy, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC.18.1.2024
Record Dates: First submitted 2024-02-07; First posted 2024-02-23 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-02

CONDITIONS: Percutaneous Nephrolithotripsy (PCNL)
MeSH Terms: interventions — Tramadol; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DP group (Active Comparator): Group I (DP group) will receive dexmedetomidine 0.5 mic/kg and paracetamol 10mg/kg
  Interventions: Drug: Dexmedetomidine 0.5 mic/kg; Drug: Paracetamol 10mg/kg
- TP group (Active Comparator): Group II (TP group) will receive tramadol 1mg/kg and paracetamol 10mg/kg.
  Interventions: Drug: Tramadol 1mg/kg; Drug: Paracetamol 10mg/kg

INTERVENTIONS:
Drug: Dexmedetomidine 0.5 mic/kg — Group I (DP group) will receive dexmedetomidine 0.5 mic/kg and paracetamol 10mg/kg,
  Arms: DP group
Drug: Tramadol 1mg/kg — Group II (TP group) will receive tramadol 1mg/kg and paracetamol 10mg/kg.
  Arms: TP group
Drug: Paracetamol 10mg/kg — Group I (DP group) will receive dexmedetomidine 0.5 mic/kg and paracetamol 10mg/kg. Group II (TP group) will receive tramadol 1mg/kg and paracetamol 10mg/kg.

SUMMARY:
The insertion of a urinary catheter in a patient undergoing a surgical procedure, especially urinary interventions, may lead to catheter-related bladder discomfort (CRBD) with varying degrees of severity during the postoperative period. Paracetamol is a drug with proven efficacy for the management of mild and moderate postoperative pain. Tramadol is a centrally acting, synthetic opioid analgesic with weak opioid agonist properties. It inhibits the detrusor activity by inhibition of type-1 muscarinic (M1) and type-3 muscarinic (M3) receptors. Dexmedetomidine, a highly selective α2-adrenergic receptor agonist, with analgesic, sedative, anxiolysis, sympatholytic, and sedative properties, is a very useful associated agent for general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age from 20 - 50 years
* ASA (The American Society of Anesthesiologists) I or II,
* undergo percutaneous nephrolithotomy (PCNL)

Exclusion Criteria:

* Patients with history of psychotic illnesses
* Opioid users
* Bladder obstruction,
* Benign prostatic hyperplasia
* Overactive bladder (OAB) defined as frequency _3 times at night or _8 times within 24 hours.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of catheter-related bladder discomfort (CRBD) | 24 hours postoperative
  The incidence of catheter-related bladder discomfort (CRBD) will be assessed at 30 minutes and 1, 2, 4, 6,8,10,12 and 24 hours postoperatively.

SECONDARY OUTCOMES:
Postoperative pain | 24 hours postoperatively
  Postoperative pain will be assessed with the Visual Analog Scale (VAS) (0, no discomfort and no pain; 10, a high level of discomfort and maximum pain)
Meperidine requirement | 24 hours postoperatively
  Total amount of consumed meperidine will be documented
Patient satisfaction | 24 hours postoperatively
  Patients' satisfaction was measured immediately postoperative and after 24 hours using a five-point Likert scale consisting of "very dissatisfied," "dissatisfied," "unsure," "satisfied," and "very satisfied.
Surgeon satisfaction | 24 hours postoperatively
  Surgeon' satisfaction was measured immediately postoperative and after 24 hours using a five-point Likert scale consisting of "very dissatisfied," "dissatisfied," "unsure," "satisfied," and "very satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Neveen Kohaf, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable request from corresponding author
Supporting Information: Study Protocol, SAP, ICF